CLINICAL TRIAL: NCT05984667
Title: C-SMART for Patients With Primary Brain Tumors: A Feasibility and Acceptability Pilot of a Novel Neuropsychological Intervention
Brief Title: C-SMART: Cognitive Strategies, Mindfulness, and Rehabilitation Therapy for Patients With Primary Brain Tumors
Acronym: C-SMART
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Psychological Foundation (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-22-20126
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Glioma, Mixed; Mild Neurocognitive Disorder; Brain Tumor
Keywords: Mindfulness; Cognitive rehabilitation; rs-fMRI
MeSH Terms: conditions — Glioma; Neurocognitive Disorders; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- C-SMART: C-SMART intervention will be provided via telehealth. Participants will complete in-person neurocognitive testing (baseline, post-intervention) as well as surveys (baseline, post-session, post-intervention) via secure email link. Exit interviews will be conducted by Zoom.
  Interventions: Behavioral: C-SMART

INTERVENTIONS:
Behavioral: C-SMART — The C-SMART intervention includes approximately 8 individual therapy sessions, each approximately 60 minutes in length, delivered weekly. C-SMART intervention components include cognitive rehabilitation and mindfulness training.

SUMMARY:
The goal of Phase IIa Trial is to determine the feasibility and acceptability of telehealth C-SMART for patients with primary brain tumor and mild neurocognitive deficits (N=36) and their caregivers (N=36) A subset (n=10) of participants will undergo rs-fMRI both pre- and post-C-SMART to test feasibility of advanced functional imaging in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed primary brain tumor diagnosis by histology or neuro-oncologist review of imaging
2. At least one domain of neurocognitive function >1.5 SD below the average or the individual's estimated premorbid functioning, using the expanded ICCTF clinical trials battery and Test of Premorbid Functioning for comparison
3. >1 month post brain surgery and/or radiation therapy, if applicable
4. Estimated premorbid intelligence >75.
5. Patients must be age 18+ and primarily English speaking

Exclusion Criteria:

1. Presence of major neurocognitive impairment that would prevent participation in the intervention, and/or severe aphasia, and/or inability to understand and provide informed consent
2. Inability to attend weekly telehealth appointments; based on EAB results
3. Clinically significant insomnia symptoms
4. < 1 month post brain surgery and/or radiation therapy
5. Unstable internet connection or an inability to work teleconferencing software. Participants will be supplied an iPad if they do not have an adequate device.
6. To participate in the fMRI portion of this study participants cannot have any metal in their bodies. For the fMRI subset, participants cannot have metal in their body as the MRI scan could cause them harm and if female of childbearing years, they cannot be pregnant as the MRI scan may pose risk to the unborn fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary brain tumor and mild neurocognitive disorder (mNCD)
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Determine feasibility of C-SMART recruitment | 10 months
  As evidenced by rates of participant screening, eligibility, and consent
Determine feasibility of C-SMART - Data collection procedures | 10 months
  As evidenced by the number of participants that complete the neurocognitive assessments pre- and post-intervention
Determine feasibility of C-SMART - Retention Rate | 11 months
  As evidenced by the number of patients that complete post-intervention measures
Determine acceptability of C-SMART intervention - Satisfaction | 10 months
  After each intervention session, participants will be sent a link for a brief post-session satisfaction survey via secure email link. In this survey, participants will rate 1) topic applicability; 2) perceived benefit of session; 3) comfort with interventionist(s); 4) overall satisfaction and 5) likelihood of recommending the program to others. Responses are ranked on a Likert-type scale from 1 being "Not at all" to 5 being "A great deal". Higher scores indicate greater satisfaction with the intervention session.
Determine acceptability of C-SMART intervention - Satisfaction - Recommendation | 10 months
  As evidenced by the number of patients that would recommend the intervention to others
Optimization of C-SMART research procedures | 8 months
  The number of participants that complete exit interviews will be audio recorded and transcribed verbatim. The PI and a second independent coder will separately review each transcript to identify common themes and develop a coding framework of free responses. All results will be reviewed for agreement and comparison to the raw data, and discrepancies will be resolved through discussion with the PI until reliability is reached (Kappa>.80)
Determine preliminary feasibility of longitudinal rs-fMRI procedures for a subset of patients | 10 months
  Completion rate of neuroimaging at post-intervention

SECONDARY OUTCOMES:
Determine feasibility of C-SMART research procedures - Patient reported outcome completion | 10 months
  Feasibility of research procedures will be assessed by the number of participants that complete the baseline survey, post-session survey, and the post-intervention survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Braun, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) to other researchers at this time.